CLINICAL TRIAL: NCT02453373
Title: Helping Stroke Patients With ThermoSuit Cooling
Acronym: SISCO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study has achieved its objectives of showing feasibility, safety, and trend for improved mRS. FDA and LRS agreed that this study should be terminated, and that a new, PIVOTAL trial should be started.
Sponsor: Life Recovery Systems (Other)
Collaborators: Tulane University School of Medicine (Other); Geisinger Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LRS-01-13-01
Record Dates: First submitted 2015-05-15; First posted 2015-05-25 (Estimated); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Stroke; Brain Ischemia
MeSH Terms: conditions — Stroke; Brain Ischemia | interventions — Magnesium Sulfate; Tissue Plasminogen Activator; Propofol; Etomidate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- ThermoSuit Cooling Induction (Experimental): Induction of therapeutic hypothermia (32-34 degrees C) using the LRS ThermoSuit System. Prior to initiating hypothermia, Magnesium Sulfate will be administered intravenously to control shivering and tPA administered intravenously (if indicated). Induction doses of propofol or etomidate will be used to aid in the suppression of patient discomfort. Neurothrombectomy will be performed if indicated.
  Interventions: Device: ThermoSuit Cooling Induction; Drug: Magnesium Sulfate; Drug: tPA; Drug: Propofol; Drug: Etomidate; Procedure: Neurothrombectomy
- Historical Control (No Intervention): Historical patients treated for ischemic stroke using conventional medical treatments, but without induced hypothermia.

INTERVENTIONS:
Device: ThermoSuit Cooling Induction — Rapid induction of therapeutic hypothermia (32-34 degrees C) using the Life Recovery Systems ThermoSuit System
  Other Names: LRS ThermoSuit
  Arms: ThermoSuit Cooling Induction
Drug: Magnesium Sulfate — Magnesium sulfate will be administered intravenously as needed to control shivering
  Other Names: Epsom salt; Magnesium sulphate
  Arms: ThermoSuit Cooling Induction
Drug: tPA — tPA will be administered intravenously if indicated
  Other Names: Tissue plasminogen activator
  Arms: ThermoSuit Cooling Induction
Drug: Propofol — Induction doses of propofol or etomidate will be used to aid in the suppression of patient discomfort
  Other Names: Diprivan
  Arms: ThermoSuit Cooling Induction
Drug: Etomidate — Induction doses of propofol or etomidate will be used to aid in the suppression of patient discomfort
  Other Names: Amidate
  Arms: ThermoSuit Cooling Induction
Procedure: Neurothrombectomy — If indicated, neurothrombectomy will be performed using an FDA-cleared device within the FDA-cleared treatment window.
  Other Names: Endovascular Thrombectomy
  Arms: ThermoSuit Cooling Induction

SUMMARY:
The aim of this study is to assess the feasibility of using the Life Recovery Systems ThermoSuit Device to induce therapeutic hypothermia (32-34°C) in victims of ischemic stroke. This feasibility clinical study will enroll a total of 30 patients with acute ischemic stroke at four clinical centers. Subjects will receive hypothermia plus conventional therapy (such as IV-tPA and/or neurothrombectomy therapies if indicated). Endpoints will include feasibility of cooling, adverse events, and neurological recovery in comparison with matched historical controls.

DETAILED DESCRIPTION:
Patients presenting to the emergency department with clinical signs and symptoms of acute ischemic stroke will undergo initial evaluation. The patient will be screened for study eligibility. A medical history and list of active medications will be documented. A physical will be conducted including the patient's temperature, hemodynamic and neurological status (NIHSS score), 12-lead ECG, and routine baseline laboratory values including magnesium, CBC, BMP, coagulation parameters, CK, CK-MB, and Troponin I. If all inclusion criteria and no exclusion criteria are present, a member of the research team will consult the patient's attending physician for permission to approach the patient. If he/she agrees, a member of the team will inform the patient or guardian about the study's purpose and obtain written informed consent. A screening log will be kept of all patients screened for this study and the reasons they were not enrolled.

Prior to initiating hypothermia, Magnesium Sulfate will be administered intravenously to control shivering and tPA administered intravenously (if indicated). Induction doses of propofol or etomidate will be used to aid in the suppression of patient discomfort. Hypothermia will generally be initiated in the ED or ICU, as soon as possible after the informed consent has been obtained. However, in cases in which neurothrombectomy is indicated and judged by the investigators to be feasible to start within 90 minutes of enrollment, cooling will be delayed until its completion, and shall afterward be initiated as soon as possible. In all cases the patient will be placed in the LRS ThermoSuit in the supine position.

Cooling will be started as specified in the Operator's Manual for the ThermoSuit device. Core temperature will be measured and monitored through a nasopharyngeal or esophageal temperature probe.

Cooling will be initiated by circulating ice-cold water (0-8°C ± 2.0°C) through the ThermoSuit, and the start time will be recorded. Patient core and TSS water temperatures will be electronically recorded. The patient will be cooled until the core temperature reaches between 32°C to 34°C. This will require approximately 5 to 20 minutes of cooling by the ThermoSuit device (not expected to be more than 30 minutes). Arterial blood pressure and heart rate will be recorded every 5 minutes from the baseline just before the start of cooling until 30 minutes after the cooling has started.

The clinician will be prompted by the automated monitor to purge the fluid from the suit when the patient's core temperature reaches approximately 33.5°C. The purging will take approximately 2 minutes. Start and stop times of purging will be recorded. The patient's body temperature should continue to decrease and then stabilize within the target range. The time at which the core temperature reaches 34°C will be recorded.

The patient will be removed from the ThermoSuit immediately after water finishes draining from the suit. The time of removal will be recorded.

Sedatives and analgesics will be administered for patient comfort as needed. Whether or not shivering occurs during cooling will be recorded, as well as start and stop times.

Body temperature will be maintained in the range of 32°C to 34°C for a period of 24 hours following the cooling induction using a cooling blanket system.

After 24 hours of therapeutic hypothermia, the patient will be re-warmed with the cooling/warming blanket until core body temperature reaches 36.5°C. This is anticipated to take approximately 8 hours.

All patients will be admitted to the intensive care unit for close monitoring of physiological parameters: blood pressure, heart rate and rhythm, arterial oxygen saturation, potassium level, acid-base balance, and indicators of infection. A head CT will be performed upon admission and 24-48 hours later. Neurological status over the first 24 hours will be closely monitored and accompanied by additional brain imaging if changes in the neurological status occur. In ICU level patients, neurological status will be evaluated q1hr with the mini-NIHSS (items 1a, 1b, 1c, and motor scores for each limb), Glasgow Coma Scale, and pupillary light response. In the case of deterioration, repeat imaging which will include CT or MRI will be performed within 48 hours to compare to admission studies. Blood pressure, heart rate and rhythm, cell count, electrolytes, magnesium, coagulation profile, cardiac enzymes, liver enzymes and serum amylase will be monitored. All neurological, cardiovascular, respiratory, digestive, hematological, and metabolic complications will be recorded and treated accordingly. Intubated patients (if any) will be extubated upon rewarming if their neurological status allows for safe extubation. NIHSS will be recorded daily, and prior to discharge.

Follow-Up on Day 5-7 post-treatment or at discharge (whichever comes first)

Records to be collected at this time will include those related to physical exam, patient temperature, hematology, clinical chemistry, ECG, blood pressure, heart rate, concomitant medications, results of any follow-up CT or MRI scans, NIHSS, Glasgow Coma Scale, pupillary light response, MRS, Quality of Life (Neuro-QOL), and any adverse events.

3 Month Follow Up

NIHSS, MRS, and Quality of Life (Neuro-QOL) will be calculated at 90 days (+/-10 days) post-stroke. Any additional adverse events will also be recorded at this time.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic cortical stroke with NIHSS > _5_;
* Treatment must be initiated within 8 hours from known time of symptom onset or, for eligible patients under the current AHA Guidelines, within the extended time window for mechanical thrombectomy of up to 24 hours.
* Patient dimension criteria: Height: 147-190 cm (58 - 75 in) Width: ≤66 cm (26 in) (elbow to elbow).

Exclusion Criteria:

* Sepsis (bacteremia and clinical syndrome within 72 h);
* Known preexisting coagulopathy, (INR > 1.3, PTT >1.5 x control), active bleeding of unknown cause, immune compromised state, thrombocytopenia (platelet count < 160,000/mm), and history of cold agglutinin disease;
* Hemodynamically significant cardiac dysrhythmias (eg. QTc interval >450 msec, bradycardia (heart rate less than 50), Mobitz Type II second degree AV block (or higher AV block), and severe ventricular dysrhythmias (sustained VT or VF) ) which cause significant hypotension (SBP ≤ 120 mmHg requiring more than two pressor medications);
* Preexistent illness with life expectancy <6 months;
* Pregnancy;
* Rapidly improving symptoms;
* Melena, or gross hematuria;
* Sickle cell disease;
* Temperature < 35°C on admission to Emergency Department;
* Recent (< 1 week) incisions;
* Any intracerebral hemorrhage;
* A history of a brain vascular lesion (e.G. aneurism or arteriovenous malformation);
* A history of brain disease or damage (e.g. neoplasm or dementia);
* Patients receiving IV tPA > 3 hours from stroke onset;
* Bradycardia (heart rate ≤ 50);
* High degree AV block;
* Ventricular tachycardia;
* Ventricular fibrillation.
* Significant hypotension < 120 mm Hg, regardless of the underlying cause

Exclusions for Patients to receive IV tPA :

* Suspicion of subarachnoid hemorrhage on pretreatment evaluation, even with normal neuroimaging;
* Systolic blood pressure greater than 185 mm of Hg or diastolic blood pressure >110 mmHg at the time of t-PA infusion and/or patient requires aggressive treatment to reduce blood pressure to within these limits;
* Seizure at onset of stroke;
* Active internal bleeding;
* Known bleeding diathesis, including but not limited to:

  * Platelet count less than 100,000/mm3
  * Heparin during the preceding 48 hours and elevated aPTT (greater than upper limit of normal for laboratory)
  * Current use of oral anticoagulants (ex: warfarin) and INR >1.7;
  * Current use of direct thrombin inhibitors or direct factor Xa inhibitors
  * Elevated prothrombin time (PT) greater than 15 seconds.
* Major surgery or other serious trauma during preceding 14 days;
* Intercranial or intraspinal surgery, stroke, serious head trauma during preceding 3 months;
* Recent arterial puncture at a non-compressible site;
* Recent lumbar puncture during preceding 7 days;
* History of intracranial hemorrhage, neoplasm, arteriovenous malformation, or aneurysm;
* Recent Acute Myocardial Infarction
* Abnormal blood glucose (<50 or >400 mg/dL)
* Suspected/confirmed endocarditis

Exclusions for Patients Receiving Neurothrombectomy >

* Patients with known hypersensitivity to nickel-titanium
* Patients with stenosis and/or pre-existing stent proximal to the thrombus site that may preclude safe recovery of the revascularization device
* Patients with angiographic evidence of carotid dissection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
Feasibility of cooling as indicated by percentage of patients cooled to target within 1 hour of start of cooling | 1 hour after start of cooling
  Feasibility of rapidly cooling victims of ischemic stroke with the ThermoSuit System to 32-34°C.
Neurological outcome as indicated by NIHSS | Hospital discharge or day 5-7 post-treatment (whichever comes first)
  NIH Stroke Scale at hospital discharge or day 5-7 post-treatment (whichever comes first)
Safety of the cooling treatment as indicated by rates of significant adverse events | 30 days
  A comparison of significant adverse event rates between the treatment and historical control group.
Neurological outcome as indicated by MRS score | Hospital discharge or day 5-7 post-treatment (whichever comes first)
  Dichotomized modified Rankin score (mRS); an mRS score of less than or equal to 2 is to be considered a good outcome
Change in neurological outcome as indicated by NIHSS | Hospital discharge or 5-7 days post-treatment (whichever comes first) and 90 +/- 10 days post-stroke
  Change in NIHSS from that measured at hospital discharge or 5-7 days post-treatment (whichever comes first) to that measured at 90 +/- 10 days post-stroke
Change in neurological status as indicated by MRS | Hospital discharge or 5-7 days post-treatment (whichever comes first) and 90 +/- 10 days post-stroke
  Change in dichotomized modified Rankin scale from that measured at hospital discharge or 5-7 days post-treatment (whichever comes first) to that measured at 90 +/- 10 days post-stroke

SECONDARY OUTCOMES:
Mortality | 90 days
  Patient death within 90 days
Quality of Life as indicated by Neuro-QOL score | Hospital discharge or 5-7 days post-treatment (whichever comes first) and 90 +/- 10 days post stroke
  Quality of Life of treated patients as assessed using Neuro-QOL forms.
Rates of procedure and device related SAEs | 0 to 90 days
  Analysis of all procedure and device related significant adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Aimee Aysenne, M.D., Principal Investigator — Tulane University
Locations (4):
- United States (4):
  - Tulane University, New Orleans, Louisiana
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - U of SC School of Medicine, Columbia, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Powers WJ, Rabinstein AA, Ackerson T, Adeoye OM, Bambakidis NC, Becker K, Biller J, Brown M, Demaerschalk BM, Hoh B, Jauch EC, Kidwell CS, Leslie-Mazwi TM, Ovbiagele B, Scott PA, Sheth KN, Southerland AM, Summers DV, Tirschwell DL; American Heart Association Stroke Council. 2018 Guidelines for the Early Management of Patients With Acute Ischemic Stroke: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2018 Mar;49(3):e46-e110. doi: 10.1161/STR.0000000000000158. Epub 2018 Jan 24. PMID 29367334
- [Derived] Salerian JA, Schock RB, Schirmer CM, Sen S, Martin-Schild S, Goren O, Kupas DF, Freedman RJ, Aysenne A. Therapeutic hypothermia with rapid thin liquid convection is safe and feasible in acute ischemic stroke patients: the SISCO pilot study. Front Neurol. 2025 Nov 7;16:1611794. doi: 10.3389/fneur.2025.1611794. eCollection 2025. PMID 41281552